CLINICAL TRIAL: NCT04597398
Title: Utility of the Evaluation of Blood Flow With Indocyanine Green in Setting the Anastomosis Site of the Remnant Esophagus in Esophagectomy With Pedicled Jejunum Reconstruction: A Case Series
Brief Title: Utility of the Evaluation of Blood Flow of the Remnant Esophagus in Esophagectomy With Pedicled Jejunum Reconstruction
Status: Completed | Type: Observational
Sponsor: Shizuoka Cancer Center (Other)
Responsible Party: Principal Investigator, Kenjiro Ishii, Doctor, Shizuoka Cancer Center
Other Study IDs: ShizuokaCC
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Esophagectomy
Keywords: Esophageal reconstructive surgery, Remnant esophagus,

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: A total of 39 patients underwent the procedure prior to June 2019
- Group B: 11 patients underwent the procedure as of June 2019
  Interventions: Device: Evaluation of blood flow with indocyanine green

INTERVENTIONS:
Device: Evaluation of blood flow with indocyanine green
  Groups: Group B

SUMMARY:
Pedicled jejunal flap can be utilized with various tips for esophageal reconstruction in patients with a history of gastrectomy, or those who have undergone synchronous esophagogastrectomy, although the rate of anastomosis leakage is high with this technique. Therefore, in the current study, we considered the utility of the evaluation of blood flow of the remnant esophagus with indocyanine green in setting the anastomosis site. We included 50 patients who underwent radical esophagectomy with pedicled jejunal flap between April 2012 and June 2020. From June 2019, the blood flow of not only the pedicled jejunum, but also the remnant esophagus were evaluated in order to set the anastomosis site of the latter because the color was not definitive criteria for judging in surgery on the remnant esophagus. Usually, the second and third jejunal vessels are transected, and if the jejunal flap cannot reach to the anastomosis point, we actively transect the marginal vessels in order to stretch the jejunal flap. Microvascular anastomosis between the jejunal branches (the second) and the internal thoracic vessels is usually made, and the anastomosis site is set at the part of the esophagus that is well-dyed with indocyanine green. A total of 39 patients underwent the procedure prior to June 2019 ( Group A), and 11 patients underwent the procedure as of June 2019 (Group B). No significant difference was found in the patients' background, type of preoperative therapy, and presence or absence of ligation of marginal vessels and two-stage operation between the two groups. Group A had 16 cases of anastomosis leakage, while Group B only has one (P < 0.05). There were no cases of significant pedicled jejunum graft necrosis. Our findings demonstrate that the evaluation of the blood flow of the remnant esophagus during setting of the anastomosis site may decrease the rate of anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent radical esophagectomy with pedicled jejunal flap between April 2012 and June 2020

Exclusion Criteria:

* patients who did not complete the esophagectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between January 2011 and June 2020, 50 patients underwent esophagectomy with pedicled jejunum reconstruction at our institute. The patients underwent subtotal esophagectomy via right thoracotomy with either an endoscopic or open procedure.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
anastomosis leakage | 1months after surgery
  the rate of anastomosis leakage between remnant esophagus and pedicled jejunum

IPD SHARING:
Plan to Share IPD: No